CLINICAL TRIAL: NCT05277090
Title: Bowel Preparation for Colonoscopy May Lead to a Higher Feasibility of Intestinal Infection: a Clinical and Basic Research
Brief Title: Bowel Preparation May Lead to a Higher Feasibility of Intestinal Infection
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yanqing Li (Other)
Responsible Party: Sponsor-Investigator, Yanqing Li, Professor, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-SDU-QILU-088
Record Dates: First submitted 2021-10-19; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Healthy
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- polyethyleneglycol only (Experimental): participants take 2L of polyethyleneglycol only
  Interventions: Drug: 2L of polyethyleneglycol
- polyethyleneglycol puls Inulin (Experimental): participants take 2L of polyethyleneglycol, subsequently take 15g inulin per day.
  Interventions: Drug: 2L of polyethyleneglycol; Dietary Supplement: inulin
- polyethyleneglycol puls probiotic combination product (Experimental): Participants take 2L of polyethyleneglycol, subsequently take 15g probiotics combination product (including Bifidobacterium lactis, Lactobacillus plantarum, inlulin, Vitamin C) per day. The probiotic combination product, named "Mei Ri Yi Jun" was produced by Wedge Pharmaceuticals.
  Interventions: Drug: 2L of polyethyleneglycol; Combination Product: probiotic combination product

INTERVENTIONS:
Drug: 2L of polyethyleneglycol — 2L of polyethyleneglycol
Dietary Supplement: inulin — 15g inulin per day
  Arms: polyethyleneglycol puls Inulin
Combination Product: probiotic combination product — participants take 2L of polyethyleneglycol, subsequently take 15g probiotics combination product (including Bifidobacterium lactis, Lactobacillus plantarum, inlulin, Vitamin C) per day. The probiotic combination product, named "Mei Ri Yi Jun" was produced by Wedge Pharmaceuticals.
  Arms: polyethyleneglycol puls probiotic combination product

SUMMARY:
An adequate bowel preparation is essential for a high quality of colonscopy. Nowdays, polyethyleneglyco is considered the most safe drug for bowel preparation, and is widely used around the world. However, previous study illustrated that bowel preparation by polyethyleneglyco could lead to qualitative changes in the intestinal microbiota both in mice and human. This study is aimed to investigate wether the changes in the intestinal microbiota could lead to a higher rate of intestinal infection.

ELIGIBILITY:
Inclusion Criteria:

* patients who agree to participant in the study

Exclusion Criteria:

* patients who couldn't stand polyethyleneglycol or inulin patients couldn't provide Informed consent patients who are suffering from sever heart disease, pulmonary disease or renal dysfunction.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Polyethyleneglycol could lead to changes in the intestinal flora | one year(from 15/3/2022 to 15/3/2023)
  People with polyethyleneglycol administration will lead to a decrease of intestinal flora quantity

SECONDARY OUTCOMES:
inulin and probiotics could improve the recovery of gut microbiota | one year(from 15/3/2022 to 15/3/2023)
  inulin and probiotics will improve the recovery of flora quantity after Polyethyleneglycol administration

CONTACTS AND LOCATIONS:
Overall Officials: Guanjun Kou, Principal Investigator — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No